CLINICAL TRIAL: NCT03564665
Title: A Randomized, Placebo Controlled, Single Blinded Trial of 400mg of Magnesium Glycinate BID Investigating the Body's Structure/Function Role of Hot Flashes.
Brief Title: Investigating Magnesium Glycinate in Structure/Function Role of Hot Flashes.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Dawn M. Mussallem, D.O., Dawn M. Mussallem, D.O., Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-000948
Record Dates: First submitted 2018-06-11; First posted 2018-06-21 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Hot Flashes
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Intervention Model Description: Randomized, Placebo Controlled, Single Blinded
Who Masked: Participant
Masking Description: Placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 400mg Magnesium Glycinate BID Arm (Experimental): Prescription for an 8 week supply (+/- 4 days) of Magnesium Glycinate will be sent to the pharmacy for patient pick up. Study Coordinator will then dispense study diaries (Supplementation Diary and Hot Flash Diary) with instructions on how to complete for the eight week study duration. Study Coordinator will discuss upcoming phone calls on Weeks 2-8 to complete the MDASI by phone and the best times to do so with the patient. Coordinator will schedule a return visit with the Patient approximately 9 weeks after the start of the study for follow-up. At follow-up, Coordinator will retrieve Patient Diaries (Hot Flash Diary and Medication Diary), perform supplement reconciliation, and exit Patient from the study.
  Interventions: Dietary Supplement: 400mg Magnesium Glycinate BID
- Control Arm (Placebo Comparator): Prescription for an 8 week supply (+/- 4 days) of placebo will be sent to the pharmacy for patient pick up. Study Coordinator will then dispense study diaries (Supplementation Diary and Hot Flash Diary) with instructions on how to complete for the eight week study duration. Study Coordinator will discuss upcoming phone calls on Weeks 2-8 to complete the MDASI by phone and the best times to do so with the patient. Coordinator will schedule a return visit with the Patient approximately 9 weeks after the start of the study for follow-up. At follow-up, Coordinator will retrieve Patient Diaries (Hot Flash Diary and Medication Diary), perform supplement reconciliation, and exit Patient from the study.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: 400mg Magnesium Glycinate BID — 400mg Magnesium Glycinate BID for 8 weeks.
  Arms: 400mg Magnesium Glycinate BID Arm
Other: Placebo — Placebo BID for 8 weeks.
  Arms: Control Arm

SUMMARY:
The goal of this study is to further evaluate the effect of magnesium on the symptoms of menopause, specifically vasomotor symptoms (VMS) in breast cancer patients and/or women at an elevated risk of breast cancer.

DETAILED DESCRIPTION:
Hot flashes are one of the most common symptoms that are experienced in women during perimenopause, menopause, and as a result of treatment of cancer such as breast cancer. Hot flashes, also known as vasomotor symptoms (VMS) may decrease a woman's quality of life due to discomfort, disruption of daily life, interruption of sleep, and worsening of depression. Previously, estrogen-based therapy was the primary treatment choice for VMS. However, in recent years, this has been considered less favorable due to the increased risk of breast cancer associated with estrogen-based therapy.

While medications such as certain antidepressants, gabapentin and clonidine are available as non-hormonal treatment options, they appear to be less effective in comparison to estrogen therapy with reported adverse effects.

Magnesium supplementation has been found to have very promising results in alleviating VMS in patients with a history of breast cancer. The goal of this study is to further investigate the effects of administering magnesium supplementation in reducing the effects of hot flashes in this targeted population. Our aim is to create a controlled trial using different dosages of magnesium glycinate in the management of hot flashes. Participants will be asked to complete surveys for data collection and analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age: 25-85 years.
* Women with a history of invasive breast cancer, DCIS, or LCIS
* Creatine labs drawn within 90 days as part of Standard of Care.
* Bothersome hot flashes (defined by their occurrence of two or more hot flashes a day and/or of sufficient severity to prompt the patient to seek therapeutic intervention).
* Presence of hot flashes for >30 days prior to study entry.
* Ability to complete questionnaire(s) by themselves or with assistance.
* Ability to provide informed written consent.
* Life expectancy ≥6 months.
* Willing to work with the enrolling institution for follow-up (during the Active Monitoring Phase of the study).
* ECOG Performance Status (PS) = 0, 1.

Exclusion Criteria:

* Pregnancy (Assessed on Intake Questionnaire. Positive Answer exclusionary)
* Any of the following current (≤4 weeks prior) or planned therapies:
* Antineoplastic chemotherapy (anti-HER2 agents allowed)
* Androgens
* Estrogens (any delivery route)
* Progestogens
* Tamoxifen, raloxifene and aromatase inhibitors are allowed, but patient must have been on a constant dose for at least 28 days and must not be expected to stop the medication during the study period
* SSRIs/SNRIs
* Gabapentin
* Clonidine
* Oxybutinin
* Stage IV or V renal disease or GFR<30 in the last 90 days

Ages: 25 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2021-04-10 (Actual); Study Completion 2021-04-10 (Actual)

PRIMARY OUTCOMES:
Percent change in hot flash frequency | 8 weeks.
  The primary endpoint of this study will be the percent change in hot flash frequency from baseline to week 8. A two independent sample z-test (assuming equal variances) or a Wilcoxon rank-sum test will be used for the analysis of this endpoint.

SECONDARY OUTCOMES:
Average change in hot flash frequency from baseline to week 8 | 8 weeks
  The secondary analysis, we will also look at the average change in hot flash frequency from baseline to week 8 and compare these means using a two-sample t-test or a Wilcoxon rank-sum test. Adverse events (as captured using the NCI CTCAE version 4) will be compared between the two investigational arms using summary statistics. Frequencies of adverse events will be compared using chi-square tests or Fisher's exact tests. Change in QOL (as measured by the MDASI) from baseline to week 8 will be compared for each question between the investigational arms using two sample t-tests or Wilcoxon rank sum tests.

CONTACTS AND LOCATIONS:
Overall Officials: Dawn M Mussallem, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

DOCUMENTS (1):
  • Study Protocol (2018-04-10): https://cdn.clinicaltrials.gov/large-docs/65/NCT03564665/Prot_000.pdf